CLINICAL TRIAL: NCT00373386
Title: Growth Hormone and Endothelial Function in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Robert Hoffman, Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Peds15
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Results first posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2017-09

CONDITIONS: Growth Hormone Deficiency; Panhypopituitarism; Short Stature
Keywords: growth hormone; endothelial function
MeSH Terms: conditions — Dwarfism, Pituitary; Combined Pituitary Hormone Deficiency; Dwarfism | interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Growth Hormone (Experimental): Growth hormone treatment 0.3 mg/kg/min
  Interventions: Drug: growth hormone

INTERVENTIONS:
Drug: growth hormone — Growth Hormone treatment

SUMMARY:
Objective: This study is designed to determine whether growth hormone treatment in children 8 to 18 years of age alters function of the lining of the arteries. This may play a role in increasing or decreasing the risk of heart disease.

Methods. Twenty children, for whom growth hormone therapy will be otherwise provided, will be studied before and 3 months after starting growth hormone. Subjects can be on other hormonal replacements but no other medications.

Each study will be done in the fasting state. The blood vessel function will be determined by measuring the change in forearm blood flow before and after blocking flow to the arm for 5 minutes. Blood will be drawn after the test to measure glucose, insulin and fats.

DETAILED DESCRIPTION:
The purpose of the research is to learn more about how the lining of arteries in the body (called the endothelium) is affected by growth hormone treatment in children and adolescents. Poor function by the blood vessels is associated with increased risk of heart disease or stroke. This research is being done because growth hormone treatment has been shown to make the endothelium work better in adults. Growth hormone treatment may have the same or different effects in children because the dose is larger in children.

Children between 8 and 18 years who are to be started on growth hormone will be eligible to participate. Blood vessel function will be studied before starting growth hormone and 3 months after. This will be done by measuring blood flow to the arm before and after 5 min of stopping blood flow to the arm. The three months of growth hormone will be given free.

ELIGIBILITY:
Inclusion Criteria:

* isolated growth hormone deficiency (peak growth hormone level less than 10 ng/ml in response to arginine-insulin stimulation with cortisol responses and thyroid function tests), panhypopituitarism with appropriate thyroxine (normal free T4 level) and cortisol replacement (8-12 mg/m2/day) and non classic growth hormone deficiency (growth velocity less than 5 cm/year; peak growth hormone >10 ng/ml).

Exclusion Criteria:

* Taking medications other than the appropriate hormonal replacement(L-thyroxine, cortisol, estrogen or testosterone, DDAVP)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2005-01; Primary Completion 2007-06 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Hoffman, MD, Study Chair — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Clinical Trials.gov

RESULTS

PARTICIPANT FLOW:
Groups:
- Growth Hormone Treatment: Growth hormone 0.3 mg/kg/week given 6 days per week
Period: Overall Study
Arm/Group | Growth Hormone Treatment
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Growth Hormone Treatment
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.9 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 9
Post occlusion forearm blood flow [Mean (Standard Deviation); unit: ml/dl*min] | 22.8 (9.9)
Glucose [Mean (Standard Deviation); unit: mg/dl] | 82 (9)
insulin [Mean (Standard Deviation); unit: uU/ml] | 5.7 (4.8)
Homa [Mean (Standard Deviation); unit: mg*uU/dl*ml] | 21 (21)
triglycerides [Mean (Standard Deviation); unit: mg/dl] | 115 (150)
ldl [Mean (Standard Deviation); unit: mg/dl] | 127 (51)
HDL [Mean (Standard Deviation); unit: mg/dl] | 44 (6)
SBP [Mean (Standard Deviation); unit: mmHg] | 96 (9)
DBP [Mean (Standard Deviation); unit: mmHg] | 47 (9)

OUTCOME MEASURES:

1. Primary Outcome: Reactive Hyperemic Response After 3 Months of Growth Hormone
Description: Forearm blood flow (FBF) was measured using strain gauge venous occlusion plethysmography using a Hokanson EC6 plethysmograph (DE Hokanson Inc, Bellevue, WA) in the left arm. With this technique sphygmomanometric cuffs were placed on the arm at the wrist and on the upper arm. During measurement the wrist cuff was inflated to 200 mmHg to occlude flow to the hand which is primarily skin blood flow and the upper arm cuff is inflated to 40 mmHG for 10 out of every 15 second to occlude venous return. FBF was obtained by measuring arm expansion with an indium-in-silastic strain gauge. Data was recorded using PowerLab and Chart 4.0 (AD Instruments, Grand Junction, CO) on a Power Mac G4 computer (Apple, Cupertino, CA).For each subject two minutes of baseline FBF were recorded and then the upper arm cuff was inflated to 200 mmHg pressure for five minutes to occlude flow to the arm. It was then released and forearm blood flow was measured for the next minute.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: ml/dl min
Groups:
- Growth Hormone Treatment: 9 subject (8 male 1 female). 8 with isolated GH deficiency (peak GH level less than 10 ng/ml in response to arginine-insulin stimulation with normal cortisol response and thyroid function tests)
  1 with panhypopitutarism on cortisol and thyroxine replacement
Arm/Group | Growth Hormone Treatment
Number analyzed (Participants) | 9
ml/dl min | 21.077 (1.937)
Statistical Analysis 1: Comparison: Growth Hormone Treatment; compared with baseline; Test type: Superiority or Other; p = 0.644, t-test, 2 sided

2. Secondary Outcome: Glucose
Description: Plasma glucose
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Growth Hormone Treatment
Number analyzed (Participants) | 9
mg/dl | 87 (9)
Statistical Analysis 1: Comparison: Growth Hormone Treatment; Compared with baseline; Test type: Superiority or Other; p = 0.018, t-test, 2 sided — Versus baseline; paired

3. Secondary Outcome: Insulin
Description: Plasma insulin
Time Frame: 3 months
Measure: Mean (Standard Error); unit: uU/ml
Arm/Group | Growth Hormone
Number analyzed (Participants) | 9
uU/ml | 11.3 (6)
Statistical Analysis 1: Comparison: Growth Hormone; Comparison to baseline; Test type: Superiority or Other; p = 0.04, t-test, 2 sided

4. Secondary Outcome: HOMA
Description: Insulin resistance
Time Frame: 3 months
Measure: Mean (Standard Error); unit: mg uU/dl ml
Groups:
- Growth Hormone Treatment: 9 subjects will have either isolated GH deficiency (peak GH level less than 10 ng/ml in response to arginine-insulin stimulation with normal cortisol response and thyroid function tests) or growth hormone deficiency with other treated pituitary deficiencies.
Arm/Group | Growth Hormone Treatment
Number analyzed (Participants) | 9
mg uU/dl ml | 43 (8)
Statistical Analysis 1: Comparison: Growth Hormone Treatment; Comparison with baseline; Test type: Superiority or Other; p = 0.004, t-test, 2 sided

5. Secondary Outcome: Triglycerides
Description: Plasma Triglycerides
Time Frame: 3 months
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Growth Hormone Treatment
Number analyzed (Participants) | 9
mg/dl | 75 (20)
Statistical Analysis 1: Comparison: Growth Hormone Treatment; Comparison with baseline; Test type: Superiority or Other; p = 0.804, t-test, 2 sided

6. Secondary Outcome: LDL
Description: LDL level
Time Frame: 3 months
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Growth Hormone Treatment
Number analyzed (Participants) | 9
mg/dl | 110 (9)
Statistical Analysis 1: Comparison: Growth Hormone Treatment; Comparison with baseline; Test type: Superiority or Other; p = 0.095, t-test, 2 sided

7. Secondary Outcome: HDL
Description: Plasma HDL
Time Frame: 3 months
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Growth Hormone Treatment
Number analyzed (Participants) | 9
mg/dl | 47 (3)
Statistical Analysis 1: Comparison: Growth Hormone Treatment; Comparison with baseline; Test type: Superiority or Other; p = 0.648, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Immediate
Arm/Group | Growth Hormone Treatment
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No